CLINICAL TRIAL: NCT04528550
Title: Intrathecal Transplantation of Autologous Bone Marrow-derived Mononuclear Cells for Treating Traumatic Acute Spinal Cord Injury
Brief Title: Autologous Bone Marrow-derived Mononuclear Cells for Acute Spinal Cord Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Xuhua Lu, Director of Traumatic Orthopaedic Department, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202082201
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: A 2:1 ratio of randomization (intervention group: control group) was used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous bone marrow-derived mononuclear cells (Experimental): Intrathecal transplantation of autologous bone marrow-derived mononuclear cells through lumbar injection in acute phase. Each included patient will receive a single dose of 100 million autologous bone marrow-derived mononuclear cells.
  Interventions: Biological: Autologous bone marrow-derived mononuclear cells
- Control (Placebo Comparator): Included patients will receive the same amount of saline through lumbar injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Autologous bone marrow-derived mononuclear cells — Intrathecal transplantation of autologous bone marrow-derived mononuclear cells through lumbar injection.
  Arms: Autologous bone marrow-derived mononuclear cells
Drug: Placebo — Included patients will receive the same amount of saline through lumbar injection.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of intrathecal transplantation of autologous bone marrow-derived mononuclear cells for the treatment of traumatic acute spinal cord injury. Spinal cord injury can be divided into three phases, which are acute (within 2 weeks), sub-acute (2 weeks to 6 months), and chronic (over 6 months). Early treatment is the key to improve the prognosis, however, the majority of clinic trails nowadays are focusing on sub-acute or chronic phase because it takes 4-6 weeks to expand the autologous stem cells. In this study, the investigators will treat patients with acute spinal cord injury with autologous bone marrow-derived mononuclear cells and compare with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 60 years
* Traumatic spinal cord injury
* ASIA Impairment Scale A-D
* The injury must be within two weeks
* Patients submitted written informed consent

Exclusion Criteria:

* Traumatic spinal cord injury with brain injury or peripheral nerve injury
* Patients with severe multiple injuries and unstable vital signs
* Non-traumatic spinal cord injury caused by spinal tumors, hematoma, myelitis, etc.
* Patients with central spinal cord injury
* Patients with a completely transected spinal cord
* Patients with fever or acute infection
* Ongoing infectious disease, such as tuberculosis, HIV, hepatitis, syphilis, etc.
* Patients with anemia, coagulopathy, and other known blood system diseases
* Patients with malignant tumour
* Patients with neurodegenerative diseases, or any neuropathies
* Patients with ankylosing spondylitis
* Patients with a previous history of spinal surgery
* Patients who are pregnant or possibly pregnant
* Patients with psychiatric, addictive or any other mental disorders that can not give a truly informed consent
* Patients who are participating in other clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
American Spinal Injury Association (ASIA) Impairment Scale | baseline, 1 month, 3 months, 6 months and 12 months post-treatment
  Change in sensory and motor function as measured by the American Spinal Injury Association (ASIA) Impairment Scale. The ASIA Impairment Scale describes a person's functional impairment (both motor and sensory) as a result of their spinal cord injury. The scale has 5 levels, ranging from A (complete) to E (normal).

SECONDARY OUTCOMES:
Incidence of adverse events | 1 month post-treatment
  Any abnormal signs, symptoms, findings, or diseases that emerge or worsen relative to baseline in 1 month post-treatment will be recorded as adverse event
Motor Evoked Potentials (MEP) and Somatosensory Evoked Potentials (SSEP) test | baseline, 3 months, 6 months and 12 months post-treatment
  Change in sensory and motor function will be measured by SSEP and MED test
Residual urine test | baseline, 3 months, 6 months and 12 months post-treatment
  Change in residual urine as measured by ultrasound test

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Lu, Principal Investigator — Shanghai Changzheng Hospotal
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided